CLINICAL TRIAL: NCT01164839
Title: Evaluation of the Factors Affecting the Diagnostic Performance of Coronary CTA With MSCT: a National Multicenter Trial
Brief Title: Evaluation of the Factors Affecting the Diagnostic Performance of Coronary Computed Tomography Angiogram (CTA) With Multi-slice Computed Tomography (MSCT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Meitan General Hospital (Unknown); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Xinan Hospital, Third Military Medical University (Unknown); Xinqiao Hospital of Chongqing (Other); Guangxi Medical University (Other); Guilin Medical College (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Chinese PLA General Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Ningxia Medical University (Other); Qinghai People's Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); RenJi Hospital (Other); Beijing Tongren Hospital (Other); The Affiliated Hospital of Tianjin Medical University (Unknown); Tang-Du Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Hospital of China Medical University (Other); Second Xiangya Hospital of Central South University (Other); Shanghai Changzheng Hospital (Other); LanZhou University (Other); Beijing Armed Police General hospital (Unknown)
Responsible Party: Kuncheng Li, Xuanwu Hospital, Capital Medical University
Other Study IDs: CCTA-CMUXW
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery; CT angiography; image quality; multicenter trial
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The multicenter study evaluates the diagnostic performance of coronary Computed Tomography Angiogram (CTA) with multi-slice computed tomography (MSCT) in comparison with X-ray coronary angiography and the factors affecting the accuracy of coronary CTA in diagnosing stenosis of coronary arteries. Furthermore, the study tends to establish the standard of image quality and associated factors that may ensure accurate diagnosis of coronary stenosis with coronary CTA.

DETAILED DESCRIPTION:
Purpose Prospectively evaluating the factors affecting the diagnostic accuracy of coronary CTA with multi-slice CT (including 64-slice CT and dual-source CT) in detecting coronary stenosis, in comparison with quantitative X-ray coronary angiography, to establish the standard of image quality and associated parameters to ensure accurate diagnosis of coronary stenosis with coronary CTA.

Detailed Description Over the past few years, the development in CT technology, especially the introduction of 64-slice multi-slice CT (64 MSCT), has permitted the application of coronary CT angiography to detect coronary stenosis in suspected patients with coronary heart diseases. Now, coronary CT angiography has been widely used worldwide. However, the accuracy of coronary CT angiography is always a concern in decision making of proper treatment, especially in determining the existence of significant stenosis in patients with visible coronary arteriosclerosis.

Factors affecting the diagnostic accuracy may include spatial resolution, temporal resolution, motion artifacts, banding artifacts, image noise level, calcification, vessel enhancement, operator dependant factors, etc. One or more factors may affect the diagnosis performance in any single case. So it is important to determine the weighting of these factors in stenosis detection and the tolerance of diagnostic accuracy to these adverse factors.

Materials and methods

1. Patient Population: About one thousand patients will be recruited over one year from our institution and other hospitals. All patients will undergo coronary CTA for suspected coronary artery disease. Then X-ray coronary angiography will be performed based on the impression on CTA findings from one radiologist (who will not participate the study) and/or clinical suspicion. Cases with both coronary CTA and X-ray coronary angiography in two weeks will be included. Our Institutional Review Board has approved the study. All patients will give informed consent. Patients with acute heart failure, severe arrhythmia and severe renal dysfunction will be excluded from cardiac studies.
2. To identify stenosis, the coronary arteries of all cases were divided into 15 segments for evaluation with coronary CTA and SCA. Coronary stenosis was recorded as percentage narrowing of lumen diameter and degree of stenosis (without stenosis, mild stenosis (≦50%), moderate stenosis (51%~75%), and severe stenosis (100%)). Experienced radiologists and cardiologists make the assessment independently in a double blind manner. The result of SCA was used as gold standard.
3. The process of coronary CTA examination of each recruited case will be carefully recorded to evaluate the factors that may affect the diagnostic performance of coronary CTA, such as heart rate, contrast injection parameters, delay time, optimal phase for reconstruction, etc. In addition, image quality will be evaluated, including the grading of motion artifact, banding artifact, enhancement, etc.
4. To evaluate operator dependant factors, all the reformations of coronary CTA will be performed by two different operators. The reformed images will also be reviewed by two different observers to evaluate the stenosis, as well as the image quality factors (motion artifacts, banding artifacts, image noise level, calcification burden, vessel enhancement).
5. Statistical analyses will be performed to evaluate the weighting of different factors in affecting the accuracy of coronary CTA.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 years to 80 years
* suspected of coronary artery disease
* capable of cooperation during coronary CT angiography
* with X-ray coronary angiography within 2 weeks after coronary CTA

Exclusion Criteria:

* refuse or not capable of signing informed consent
* pregnant or nursing period
* acute heart failure
* severe arrhythmia
* allergic to iodine
* severe renal failure
* not capable of breathholding
* acute myocardial infarction or previous myocardial infarction
* previous stent implantation
* change of clinical status between coronary CTA and X-ray coronary angiography

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive eligible patients who undergo both coronary CTA and X-ray coronary angiography
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kuncheng Li, MD, PhD, Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China